CLINICAL TRIAL: NCT02592876
Title: A Randomized, Open-Label Phase 2 Study of Denintuzumab Mafodotin (SGN-CD19A) Plus Rituximab, Ifosfamide, Carboplatin, and Etoposide (19A+RICE) Chemotherapy vs. RICE in the Treatment of Patients With Relapsed or Refractory Diffuse Large B-Cell Lymphoma (DLBCL) Who Are Candidates for Autologous Stem Cell Transplant
Brief Title: Treatment Study of Denintuzumab Mafodotin (SGN-CD19A) Plus RICE Versus RICE Alone for Diffuse Large B-Cell Lymphoma
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: Sponsor decision based on portfolio prioritization
Sponsor: Seagen Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: SGN19A-003
Record Dates: First submitted 2015-10-29; First posted 2015-10-30 (Estimated); Results first posted 2019-05-17 (Actual); Last update posted 2019-05-17 (Actual); Status verified 2019-04

CONDITIONS: Lymphoma, B-cell; Lymphoma, Large B-Cell, Diffuse; Lymphoma, Follicular, Grade 3b; Follicular Lymphoma, Grade 3b
Keywords: Antibodies, Monoclonal; Antibody-Drug Conjugate; Antigens, CD19; Autologous Stem Cell Transplant; Drug Therapy; Follicular Lymphoma Grade 3b; Hematologic Diseases; Immune System Diseases; Immunoproliferative Disorders; Immunotherapy; Lymphatic Diseases; Lymphoma; Lymphoma, B-Cell; Lymphoma, Large B-Cell, Diffuse; Lymphoma, Non-Hodgkin; Monomethylauristatin F; Neoplasms; Neoplasms by Histologic Type; Transformed Lymphoma / DLBCL; Rituximab; Ifosfamide; Carboplatin; Etoposide
MeSH Terms: conditions — Lymphoma, B-Cell; Lymphoma, Large B-Cell, Diffuse; Lymphoma; Lymphoma, Follicular; Hematologic Diseases; Immune System Diseases; Immunoproliferative Disorders; Lymphatic Diseases; Lymphoma, Non-Hodgkin; Neoplasms; Neoplasms by Histologic Type | interventions — Rituximab; Ifosfamide; Carboplatin; Etoposide

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- 19A+RICE (Experimental): Denintuzumab mafodotin plus rituximab, ifosfamide, carboplatin, and etoposide
  Interventions: Drug: denintuzumab mafodotin; Drug: rituximab; Drug: ifosfamide; Drug: carboplatin; Drug: etoposide
- RICE (Active Comparator): Rituximab, ifosfamide, carboplatin, and etoposide
  Interventions: Drug: rituximab; Drug: ifosfamide; Drug: carboplatin; Drug: etoposide

INTERVENTIONS:
Drug: denintuzumab mafodotin — Denintuzumab mafodotin 3 mg/kg by intravenous (IV) infusion, every 3 weeks for up to 3 cycles.
  Other Names: SGN-CD19A
  Arms: 19A+RICE
Drug: rituximab — 375 mg/m^2 by IV infusion, every 3 weeks for up to 3 cycles
Drug: ifosfamide — 5000 mg/m^2 by IV infusion over a 24-hour period, every 3 weeks for up to 3 cycles
Drug: carboplatin — AUC 5mg/mL x min by IV infusion, every 3 weeks for up to 3 cycles
Drug: etoposide — 100 mg/m^2 per day by IV infusion for 3 days, every 3 weeks for up to 3 cycles

SUMMARY:
The purpose of this randomized, open-label study is to evaluate the safety and efficacy of denintuzumab mafodotin plus RICE (rituximab, ifosfamide, carboplatin, and etoposide) when compared to RICE alone in the treatment of patients with relapsed or refractory diffuse large B-cell lymphoma (DLBCL) or Grade 3b follicular lymphoma. Eligible patients must also be candidates for autologous stem cell transplant. Patients will be randomly assigned in a 1:1 ratio to receive 3 cycles of study treatment with either denintuzumab mafodotin + RICE or RICE alone. The study will assess whether there is a difference between the 2 groups in the side effects that are reported and the number of patients who achieve complete remission at the end of their study treatment.

ELIGIBILITY:
Inclusion Criteria:

* Pathologically confirmed diagnosis of relapsed or refractory diffuse large B-cell lymphoma (DLBCL; including de novo and transformed DLBCL) or Grade 3b follicular lymphoma
* Available representative tissue from the most recent biopsy after the last therapy; if such tissue is not available, a fresh biopsy must be obtained
* Received only frontline CD20-directed immunotherapy with anthracycline- or anthracenedione-based multi-agent chemotherapy. Monotherapy rituximab or other CD20-directed immunotherapy as maintenance therapy prior to frontline chemotherapy, and radiotherapy in a limited field or as part of the frontline treatment plan are permitted.
* Achieved a response of stable disease, partial response, or complete response following the last cycle of frontline treatment. In addition, patients must have relapsed less than or equal to 6 months from the completion of frontline therapy at the time of initial dosing in this clinical trial.
* Considered eligible for high-dose chemotherapy followed by autologous stem cell transplant (ASCT)
* Fluorodeoxyglucose (FDG)-avid disease by positive emission tomography (PET), and measurable disease greater than 1.5 cm in diameter
* Eastern Cooperative Oncology Group (ECOG) performance less than or equal to 2
* Adequate kidney and hematologic function assessed from baseline laboratory data

Exclusion Criteria:

* Previous history of indolent lymphoma treated with more than 1 multi-agent chemotherapy regimen or previous cancer therapy for recurrent DLBCL or Grade 3b follicular lymphoma
* History of autologous or allogeneic stem cell transplant
* History of another primary invasive cancer, hematologic malignancy, or myelodysplastic syndrome that has not been in remission for at least 1 year
* History of progressive multifocal leukoencephalopathy (PML)
* Cerebral/meningeal disease related to the underlying malignancy that has not been definitively treated
* Known urinary tract obstruction
* Patients with the following ocular conditions: corneal disorders, monocular vision (i.e., best corrected visual acuity greater than or equal to 20/200 in one eye), or active ocular disorders requiring treatment

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 81 (Actual)
Dates: Start 2015-10 (Actual); Primary Completion 2018-04-20 (Actual); Study Completion 2018-04-20 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Juan Pinelli, PA-C, MMSc, Study Director — Seagen Inc.
Locations (29):
- United States (29):
  - University of Arkansas for Medical Sciences, Little Rock, Arkansas
  - City of Hope National Medical Center, Duarte, California
  - Scripps Mercy Cancer Center, San Diego, California
  - Colorado Blood Cancer Institute, Denver, Colorado
  - Yale Cancer Center, New Haven, Connecticut
  - Shands Cancer Center / University of Florida, Gainesville, Florida
  - University of Miami, Miami, Florida
  - H. Lee Moffitt Cancer Center & Research Institute, Tampa, Florida
  - Winship Cancer Institute / Emory University School of Medicine, Atlanta, Georgia
  - Rush University Medical Center, Chicago, Illinois
  - University of Chicago, Chicago, Illinois
  - Cardinal Bernardin Cancer Center / Loyola University Medical Center, Maywood, Illinois
  - University of Kansas Cancer Center, Westwood, Kansas
  - Beth Israel Deaconess Medical Center, Boston, Massachusetts
  - Dana Farber Cancer Institute, Boston, Massachusetts
  - University of Minnesota, Minneapolis, Minnesota
  - Washington University School of Medicine, St Louis, Missouri
  - Hackensack University Medical Center, Hackensack, New Jersey
  - University of New Mexico Cancer Center, Albuquerque, New Mexico
  - Memorial Sloan Kettering Cancer Center, New York, New York
  - UNC Lineberger Comprehensive Cancer Center / University of North Carolina, Chapel Hill, North Carolina
  - Levine Cancer Institute, Charlotte, North Carolina
  - Duke University Medical Center, Durham, North Carolina
  - MD Anderson Cancer Center / University of Texas, Houston, Texas
  - San Antonio Military Medical Center, San Antonio, Texas
  - University of Virginia, Charlottesville, Virginia
  - Seattle Cancer Care Alliance / University of Washington, Seattle, Washington
  - Carbone Cancer Center / University of Wisconsin, Madison, Wisconsin
  - Medical College of Wisconsin (Milwaukee), Milwaukee, Wisconsin

RESULTS

PARTICIPANT FLOW:
Groups:
- RICE: Rituximab, ifosfamide, carboplatin, and etoposide
  rituximab: 375 mg/m2 by IV infusion, every 3 weeks for up to 3 cycles
  ifosfamide: 5000 mg/m2 by IV infusion over a 24-hour period, every 3 weeks for up to 3 cycles
  carboplatin: AUC 5 by IV infusion, every 3 weeks for up to 3 cycles
  etoposide: 100 mg/m2 per day by IV infusion for 3 days, every 3 weeks for up to 3 cycles
- 19A+RICE: Denintuzumab mafodotin plus rituximab, ifosfamide, carboplatin, and etoposide
  denintuzumab mafodotin: Denintuzumab mafodotin 3 mg/kg by intravenous (IV) infusion, every 3 weeks for up to 3 cycles.
  rituximab: 375 mg/m2 by IV infusion, every 3 weeks for up to 3 cycles
  ifosfamide: 5000 mg/m2 by IV infusion over a 24-hour period, every 3 weeks for up to 3 cycles
  carboplatin: AUC 5 by IV infusion, every 3 weeks for up to 3 cycles
  etoposide: 100 mg/m2 per day by IV infusion for 3 days, every 3 weeks for up to 3 cycles
Period: Overall Study
Arm/Group | RICE | 19A+RICE
Started | 41 | 40
Received Study Drug | 40 | 40
Completed Treatment | 34 | 32
Completed | 0 | 0
Not Completed | 41 | 40
Not completed — Withdrawal by Subject | 3 | 3
Not completed — Study Termination by Sponsor | 32 | 27
Not completed — Lost to Follow-up | 0 | 1
Not completed — Death | 6 | 9

BASELINE CHARACTERISTICS:
Population: Includes all randomized participants
Groups:
- Total: Total of all reporting groups
Arm/Group | RICE | 19A+RICE | Total
Number analyzed (Participants) | 41 | 40 | 81
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 28 | 24 | 52
  >=65 years | 13 | 16 | 29
Age, Continuous [Median (Full Range); unit: years] | 60.0 [25 to 74] | 62.5 [20 to 76] | 61.0 [20 to 76]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 16 | 13 | 29
  Male | 25 | 27 | 52
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 3 | 5 | 8
  Not Hispanic or Latino | 37 | 35 | 72
  Unknown or Not Reported | 1 | 0 | 1
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 1 | 1 | 2
  Native Hawaiian or Other Pacific Islander | 1 | 0 | 1
  Black or African American | 1 | 1 | 2
  White | 37 | 36 | 73
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 1 | 2 | 3
Region of Enrollment [Number; unit: participants]
  United States | 41 | 40 | 81
Eastern Cooperative Oncology Group (ECOG) Performance Status [Count of Participants; unit: Participants] — 0=Normal activity; 1=Symptoms but ambulatory; 2=In bed <50% of the time; 3= In bed >50% of the time; 4=100% bedridden; 5=Dead
  Participants
    Grade 0 | 17 | 19 | 36
    Grade 1 | 21 | 21 | 42
    Grade 2 | 3 | 0 | 3

OUTCOME MEASURES:

1. Primary Outcome: Complete Remission Rate Per Independent Review Facility
Description: Number of patients with complete metabolic response by PET (positive emission tomography) and CT (computed tomography) scans, or complete radiologic response by CT only.
Time Frame: Up to 4 months
Population: The modified Intent-to-Treat (mITT) analysis set includes all patients who were randomized to the recommended dose level of 19A+RICE or RICE and received at least 1 cycle of study treatment.
Measure: Count of Participants; unit: Participants
Arm/Group | RICE | 19A+RICE
Number analyzed (Participants) | 40 | 40
Participants | 18 | 25

2. Secondary Outcome: Number of Participants With Adverse Events (AEs)
Description: Treatment-emergent adverse events (TEAEs) are presented and defined as newly occurring (not present at baseline) or worsening after first dose of investigational product. AE severity and seriousness are assessed independently. 'Severity' characterizes the intensity of an AE and is graded using the National Cancer Institute's Common Terminology Criteria for Adverse Events (NCI CTCAE), version 4.03. An AE is considered 'serious' if it is life-threatening, fatal, requires hospitalization, or is otherwise considered to be medically significant.
Time Frame: Up to 4 months
Population: The safety analysis set includes all patients who received any amount of denintuzumab mafodotin or any component of RICE. Treatment group is determined using the actual treatment arm received, regardless of the randomization treatment assignment.
Measure: Count of Participants; unit: Participants
Arm/Group | RICE | 19A+RICE
Number analyzed (Participants) | 40 | 40
Participants
  Treatment-emergent AE (TEAE) | 39 | 40
  Treatment-related AEs | 38 | 40
  Grade 3 or Higher TEAEs | 31 | 38
  Serious AEs (SAEs) | 13 | 19
  Treatment-related SAEs | 9 | 13
  AEs Leading to Dose Delay | 3 | 8
  AEs Leading to Dose Reduction | 3 | 5
  AEs Leading to Treatment Discontinuation | 2 | 3

3. Secondary Outcome: Number of Participants With Laboratory Abnormalities
Description: Number of participants who experienced a maximum post-baseline laboratory toxicity of Grade 3 or higher (per National Cancer Institute's Common Terminology Criteria for Adverse Events, version 4.03).
Time Frame: Up to 4 months
Population: as for outcome 2
Measure: Count of Participants; unit: Participants
Arm/Group | RICE | 19A+RICE
Number analyzed (Participants) | 40 | 40
Participants
  Any Hematology Test | 37 | 37
  Hemoglobin Low | 19 | 18
  Leukocytes High | 1 | 0
  Leukocytes Low | 23 | 24
  Lymphocytes High | 2 | 0
  Lymphocytes Low | 34 | 31
  Neutrophils Low | 22 | 22
  Platelets Low | 26 | 35
  Any Chemistry Test | 18 | 16
  Alanine Aminotransferase High | 3 | 3
  Aspartate Aminotransferase High | 1 | 2
  Calcium High | 4 | 0
  Calcium Low | 0 | 2
  Creatinine High | 0 | 1
  Glucose High | 4 | 3
  Phosphate Low | 9 | 8
  Potassium Low | 3 | 5
  Sodium Low | 4 | 3
  Urate High | 2 | 0

4. Secondary Outcome: Objective Response Rate (ORR)
Description: ORR is defined as the proportion of patients with complete remission (CR) or partial remission (PR) per independent review facility (IRF) at the end of treatment.
Time Frame: Up to 4 months
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | RICE | 19A+RICE
Number analyzed (Participants) | 40 | 40
Participants | 30 | 32

5. Secondary Outcome: Duration of Complete Response (CR)
Description: Defined as the time from the start of the first radiographic documentation of CR per investigator to the first documentation of progressive disease, death due to any cause, or receipt of subsequent anticancer therapy, whichever comes first.
Time Frame: Up to 27.9 months
Population: as for outcome 1
Measure: Median (Inter-Quartile Range); unit: months
Arm/Group | RICE | 19A+RICE
Number analyzed (Participants) | 40 | 40
months | NA [NA to NA] — Insufficient number of events observed | NA [NA to NA] — Insufficient number of events observed

6. Secondary Outcome: Duration of Objective Response (OR)
Description: Duration of OR is defined as the time from the start of the first radiographic documentation of OR per investigator to the first documentation of PD, death due to any cause, or receipt of subsequent anticancer therapy, whichever comes first.
Time Frame: Up to 27.9 months
Measure: Median (Inter-Quartile Range); unit: months
Arm/Group | RICE | 19A+RICE
Number analyzed (Participants) | 40 | 40
months | NA [8.15 to NA] — Insufficient number of events observed | NA [NA to NA] — Insufficient number of events observed

7. Secondary Outcome: Progression-free Survival (PFS)
Description: PFS is defined as the time from randomization to first documentation of disease progression per investigator, death due to any cause, or receipt of subsequent anticancer therapy, whichever comes first.
Time Frame: Up to 30 months
Population: as for outcome 1
Measure: Median (Inter-Quartile Range); unit: months
Arm/Group | RICE | 19A+RICE
Number analyzed (Participants) | 40 | 40
months | NA [2.86 to NA] — Insufficient number of events observed | NA [5.82 to NA] — Insufficient number of events observed

8. Secondary Outcome: Overall Survival (OS)
Description: OS is defined as the time from date of randomization to date of death due to any cause. In the absence of confirmation of death, survival time will be censored at the last date the patient is known to be alive.
Time Frame: Up to 30 months
Population: as for outcome 1
Measure: Median (Inter-Quartile Range); unit: months
Arm/Group | RICE | 19A+RICE
Number analyzed (Participants) | 40 | 40
months | NA [NA to NA] — Insufficient number of events observed | NA [10.97 to NA] — Insufficient number of events observed

9. Secondary Outcome: Number of Patients Achieving Peripheral Blood Stem Cell (PBSC) Mobilization
Description: Defined as the number of patients who are able to adequately mobilize PBSC per investigator assessment on or after completion of study treatment, prior to subsequent anticancer therapy.
Time Frame: Up to 30 months
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | RICE | 19A+RICE
Number analyzed (Participants) | 40 | 40
Participants
  Patients with attempted stem cell collection(s) | 28 | 24
  Patients with sufficient stem cell collection | 26 | 21

10. Secondary Outcome: Number of Patients Receiving Autologous Stem Cell Transplant (ASCT)
Description: Number of patients receiving ASCT after completion of study treatment (EOT), prior to subsequent anticancer therapy.
Time Frame: Up to 30 months
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | RICE | 19A+RICE
Number analyzed (Participants) | 40 | 40
Participants
  Patients planned to receive ASCT at EOT | 28 | 25
  Patients who received ASCT at EOT | 25 | 22

ADVERSE EVENTS:
Time Frame: Up to 30 months
Arm/Group | RICE | 19A+RICE
All-Cause Mortality (participants affected / at risk) | 6/40 | 9/40
Serious Adverse Events (participants affected / at risk) | 13/40 | 19/40
Other Adverse Events (participants affected / at risk) | 40/40 | 40/40
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | RICE (N=40) | 19A+RICE (N=40)
Anaemia (Blood and lymphatic system disorders) | 0 | 3
Febrile neutropenia (Blood and lymphatic system disorders) | 6 | 8
Thrombocytopenia (Blood and lymphatic system disorders) | 1 | 1
Tachycardia (Cardiac disorders) | 1 | 0
Gastric haemorrhage (Gastrointestinal disorders) | 0 | 1
Gastritis (Gastrointestinal disorders) | 0 | 1
Gastrointestinal haemorrhage (Gastrointestinal disorders) | 0 | 1
Intestinal fistula (Gastrointestinal disorders) | 0 | 1
Intestinal obstruction (Gastrointestinal disorders) | 0 | 1
Nausea (Gastrointestinal disorders) | 0 | 1
Pancreatitis (Gastrointestinal disorders) | 0 | 1
Pancreatitis acute (Gastrointestinal disorders) | 0 | 1
Rectal haemorrhage (Gastrointestinal disorders) | 0 | 1
Small intestinal obstruction (Gastrointestinal disorders) | 0 | 1
Vomiting (Gastrointestinal disorders) | 0 | 1
Pyrexia (General disorders) | 1 | 1
External ear cellulitis (Infections and infestations) | 1 | 0
Lung infection (Infections and infestations) | 0 | 1
Otitis externa (Infections and infestations) | 1 | 0
Pneumonia (Infections and infestations) | 1 | 0
Rhinovirus infection (Infections and infestations) | 0 | 1
Sepsis (Infections and infestations) | 0 | 1
Septic shock (Infections and infestations) | 0 | 1
Gastrointestinal stoma complication (Injury, poisoning and procedural complications) | 1 | 0
Hip fracture (Injury, poisoning and procedural complications) | 1 | 0
Post procedural haemorrhage (Injury, poisoning and procedural complications) | 0 | 1
Toxicity to various agents (Injury, poisoning and procedural complications) | 1 | 0
Transfusion reaction (Injury, poisoning and procedural complications) | 0 | 1
Alanine aminotransferase increased (Investigations) | 0 | 1
Aspartate aminotransferase increased (Investigations) | 0 | 1
Hepatic enzyme increased (Investigations) | 1 | 0
Platelet count decreased (Investigations) | 0 | 3
White blood cell count decreased (Investigations) | 0 | 2
Hypokalaemia (Metabolism and nutrition disorders) | 0 | 1
Malignant pleural effusion (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Depressed level of consciousness (Nervous system disorders) | 1 | 0
Headache (Nervous system disorders) | 0 | 1
Neurotoxicity (Nervous system disorders) | 0 | 1
Syncope (Nervous system disorders) | 0 | 1
Acute kidney injury (Renal and urinary disorders) | 1 | 0
Acute respiratory failure (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Haemothorax (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Mediastinal mass (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Pruritus (Skin and subcutaneous tissue disorders) | 0 | 1
Urticaria (Skin and subcutaneous tissue disorders) | 0 | 1
Hypotension (Vascular disorders) | 1 | 0
Orthostatic hypotension (Vascular disorders) | 0 | 1
Vena cava thrombosis (Vascular disorders) | 1 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | RICE (N=40) | 19A+RICE (N=40)
Anaemia (Blood and lymphatic system disorders) | 23 | 19
Neutropenia (Blood and lymphatic system disorders) | 3 | 9
Thrombocytopenia (Blood and lymphatic system disorders) | 15 | 23
Dry eye (Eye disorders) | 4 | 10
Foreign body sensation in eyes (Eye disorders) | 0 | 4
Keratitis (Eye disorders) | 0 | 4
Keratopathy (Eye disorders) | 3 | 27
Photophobia (Eye disorders) | 1 | 8
Vision blurred (Eye disorders) | 5 | 26
Abdominal pain (Gastrointestinal disorders) | 1 | 5
Constipation (Gastrointestinal disorders) | 11 | 12
Diarrhoea (Gastrointestinal disorders) | 5 | 9
Dry mouth (Gastrointestinal disorders) | 3 | 1
Dyspepsia (Gastrointestinal disorders) | 3 | 2
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 3 | 1
Nausea (Gastrointestinal disorders) | 25 | 26
Stomatitis (Gastrointestinal disorders) | 2 | 2
Vomiting (Gastrointestinal disorders) | 11 | 12
Asthenia (General disorders) | 2 | 3
Chills (General disorders) | 5 | 5
Fatigue (General disorders) | 21 | 19
Oedema peripheral (General disorders) | 7 | 5
Pyrexia (General disorders) | 4 | 4
Contusion (Injury, poisoning and procedural complications) | 2 | 3
Alanine aminotransferase increased (Investigations) | 2 | 2
Aspartate aminotransferase increased (Investigations) | 2 | 3
Blood creatinine increased (Investigations) | 3 | 1
Platelet count decreased (Investigations) | 0 | 6
Weight decreased (Investigations) | 2 | 2
Decreased appetite (Metabolism and nutrition disorders) | 8 | 7
Dehydration (Metabolism and nutrition disorders) | 3 | 3
Hyperglycaemia (Metabolism and nutrition disorders) | 3 | 3
Hypokalaemia (Metabolism and nutrition disorders) | 6 | 7
Hypomagnesaemia (Metabolism and nutrition disorders) | 8 | 7
Hyponatraemia (Metabolism and nutrition disorders) | 1 | 3
Hypophosphataemia (Metabolism and nutrition disorders) | 3 | 3
Back pain (Musculoskeletal and connective tissue disorders) | 1 | 3
Bone pain (Musculoskeletal and connective tissue disorders) | 4 | 0
Pain in extremity (Musculoskeletal and connective tissue disorders) | 1 | 3
Dizziness (Nervous system disorders) | 5 | 6
Dysgeusia (Nervous system disorders) | 3 | 2
Headache (Nervous system disorders) | 7 | 9
Paraesthesia (Nervous system disorders) | 0 | 4
Peripheral sensory neuropathy (Nervous system disorders) | 4 | 0
Syncope (Nervous system disorders) | 3 | 2
Insomnia (Psychiatric disorders) | 3 | 6
Dysuria (Renal and urinary disorders) | 3 | 1
Cough (Respiratory, thoracic and mediastinal disorders) | 2 | 6
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 7 | 3
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 3 | 4
Hiccups (Respiratory, thoracic and mediastinal disorders) | 4 | 6
Alopecia (Skin and subcutaneous tissue disorders) | 5 | 7
Night sweats (Skin and subcutaneous tissue disorders) | 2 | 3
Hypotension (Vascular disorders) | 2 | 2

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes

DOCUMENTS (2):
  • Study Protocol (2017-10-28): https://cdn.clinicaltrials.gov/large-docs/76/NCT02592876/Prot_000.pdf
  • Statistical Analysis Plan (2016-10-21): https://cdn.clinicaltrials.gov/large-docs/76/NCT02592876/SAP_001.pdf